CLINICAL TRIAL: NCT04715516
Title: A Brief Intervention to Increase Knowledge of Alcohol as a Breast Cancer Risk Factor Among Women Attending Breast Screening Services (Health4Her): A Pilot Randomised Controlled Trial
Brief Title: Increasing Knowledge of Alcohol as a Risk Factor for Breast Cancer Among Women Attending Breast Screening Services
Acronym: Health4Her
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turning Point (Other)
Collaborators: Eastern Health (Other); Monash University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: LR19/011/50551
Record Dates: First submitted 2021-01-11; First posted 2021-01-20 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Health Knowledge, Attitudes, Practice; Alcohol Consumption
Keywords: Women's health; Public Health; Health promotion/education
MeSH Terms: conditions — Behavior; Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- alcohol brief intervention + lifestyle health promotion (Experimental): The intervention arm will receive 4 minutes of alcohol brief intervention, and 3 minutes of lifestyle health promotion (physical activity; maintaining a healthy weight), to increase knowledge of how to improve women's health and reduce breast cancer risk. Alcohol and lifestyle information will be delivered by way of an animation on an iPad. Participant responses to questions about current alcohol use will branch to personalised feedback consistent with level of alcohol consumption (i.e. drinking within or above current Australian Alcohol Guidelines).
  Take-home pamphlets - a pamphlet summarising the alcohol information presented during the animation, and a pamphlet on nutrition to maintain a healthy weight, will be provided.
  Interventions: Behavioral: alcohol brief intervention; Behavioral: lifestyle health promotion
- lifestyle health promotion, not inclusive of alcohol information (Other): The control arm will receive 3 minutes of lifestyle health promotion (physical activity; maintaining a healthy weight) to increase knowledge of how to improve women's health and reduce breast cancer risk, not inclusive of alcohol information. Lifestyle information will be delivered by way of an animation on an iPad.
  Take-home pamphlet - a pamphlet on nutrition to maintain a healthy weight will be provided.
  Interventions: Behavioral: lifestyle health promotion

INTERVENTIONS:
Behavioral: alcohol brief intervention — Nested within the lifestyle health promotion provided in both conditions, participants randomised to the experimental condition will receive an alcohol brief intervention. The strong evidence-base for alcohol brief intervention, amplified by Co-Investigators' Smith and Bragge's (BehaviourWorks) approaches to applied behaviour change, has provided the framework for the development of the alcohol brief intervention used in this study. This intervention comprises personalised feedback on alcohol consumption levels, comparison to gender/age drinking norms, and information and behaviour-change content regarding alcohol consumption (i.e. negative-framed messaging around alcohol risks and harms, positive-framed messaging on the health benefits of reducing alcohol intake, alcohol harm reduction strategies).
  Arms: alcohol brief intervention + lifestyle health promotion
Behavioral: lifestyle health promotion — Lifestyle health promotion specific to physical activity and maintaining a healthy weight, developed to be relevant to women attending breast screening services, will be provided.

SUMMARY:
Alcohol is a major modifiable risk factor for breast cancer in women, yet this is not widely understood by health practitioners or policy makers, let alone the general population. The investigators aim to test the effects of a targeted alcohol and lifestyle brief intervention for women attending breast screening services, to improve knowledge of alcohol as a risk factor for breast cancer and reduce harmful alcohol use.

ELIGIBILITY:
Inclusion Criteria:

* female
* attending breast screening service for a routine mammography
* 40-74 years
* English as a first language or fluent
* regular access to a telephone
* able to provide informed consent to participate
* any level of alcohol consumption (including non-drinkers)

Exclusion Criteria:

* hearing impairment sufficient to prohibit a telephone interview
* pregnancy
* not able to read or comprehend English to provide informed consent or receive the brief intervention

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Knowledge of alcohol as a breast cancer risk factor | 4-weeks post-randomisation
  Proportion of participants accurately identifying alcohol as a clear risk factor for breast cancer

SECONDARY OUTCOMES:
Drinking within current Australian Alcohol Guidelines | 4-weeks and 3-months post-randomisation
  Proportion of participants drinking less than or equal to 10 standard drinks per week (within current Australian Alcohol Guidelines) (14-day Timeline Followback, TLFB)
Drinking within current Australian Alcohol Guidelines (among participants who drink more than 10 standard drinks per week) | 4-weeks and 3-months post-randomisation
  Among participants who drink more than 10 standard drinks per week at baseline: Proportion of participants drinking less than or equal to 10 standard drinks per week. (14-day TLFB)
Alcohol consumption | 4-weeks and 3-months post-randomisation
  Change in alcohol consumption (14-day TLFB; AIHW alcohol frequency quantity items)
Alcohol consumption (among participants who drink more than 10 standard drinks per week) | 4-weeks and 3-months post-randomisation
  Among participants who drink more than 10 standard drinks per week at baseline: Change in alcohol consumption (14-day TLFB; AIHW alcohol frequency quantity items)
Health literacy - attitudes | 4-weeks post-randomisation
  Change in participants' attitudes regarding alcohol and breast cancer risk (5-point scale, strongly agree to strongly disagree; items adapted from previous literature, e.g. Fisher et al. 2017)
Health literacy - knowledge | 4-weeks post-randomisation
  Proportion of participants accurately identifying i) the amount of alcohol in an Australian standard drink; ii) the number of standard drinks in an average restaurant serve of red wine; iii) the maximum number of standard drinks per week recommended by current Australian Alcohol Guidelines (multiple choice and open-ended questions, adapted from previous literature, e.g. Bowden et al. 2014)
Health literacy - access to health information | 4-weeks post-randomisation
  Proportion of participants who have accessed health information on i) alcohol harms, ii) alcohol and breast cancer risk, and iii) alcohol harm-reduction
General health | 4-weeks and 3-months post-randomisation
  Change in general health (SF-12)
Quality of life | 4-weeks and 3-months post-randomisation
  Change in quality of life (EUROHIS-QOL single item)

OTHER OUTCOMES:
Program evaluation | Through study completion, approximately 9 months
  Mixed-methods program evaluation (Glasgow et al.'s RE-AIM framework)

CONTACTS AND LOCATIONS:
Overall Officials: Dan I Lubman, Principal Investigator — Turning Point, Eastern Health; Monash University
Locations (1):
- Maroondah BreastScreen, Ringwood East, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
We do not have Ethics approval to seek patient permission to share data outside this study, other than for related projects conducted by the research team.

REFERENCES:
- [Derived] Grigg J, Manning V, Lockie D, Giles M, Bell RJ, Stragalinos P, Bernard C, Greenwood CJ, Volpe I, Smith L, Bragge P, Lubman DI. A brief intervention for improving alcohol literacy and reducing harmful alcohol use by women attending a breast screening service: a randomised controlled trial. Med J Aust. 2023 Jun 19;218(11):511-519. doi: 10.5694/mja2.51991. Epub 2023 May 29. PMID 37247850
- [Derived] Grigg J, Manning V, Lockie D, Giles M, Bell R, Stragalinos P, Bernard C, Volpe I, Greenwood CJ, Smith L, Bragge P, Lubman DI. A Brief Intervention for Improving Alcohol Literacy and Addressing Harmful Alcohol Use Among Women Attending an Australian Breast Screening Service (Health4her): Protocol for a Hybrid Effectiveness-Implementation Trial. JMIR Res Protoc. 2023 Mar 30;12:e44867. doi: 10.2196/44867. PMID 36995739

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Brief overview (2021-08-08): https://cdn.clinicaltrials.gov/large-docs/16/NCT04715516/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Full SAP (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/16/NCT04715516/SAP_001.pdf